CLINICAL TRIAL: NCT02335606
Title: Real World Effectiveness of Abatacept in Rheumatoid Arthritis Patients: a Prospective, Single-arm, Multi-center Observational Study in Taiwan
Brief Title: Real World Effectiveness of Abatacept in Rheumatoid Arthritis Patients: a Prospective, Single-arm, Open-label, Multi-center Observational Study in Taiwan
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM101-440
Record Dates: First submitted 2015-01-07; First posted 2015-01-12 (Estimated); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients treating with Abatacept: Patients who are abatacept naive and are initiating abatacept treatment (either IV or SC) including those that are switching from another bDMARD, as well as, patients currently being treated with IV or SC abatacept some of which may have switched from IV abatacept to SC abatacept

SUMMARY:
Abatacept Registry in Taiwan

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* ≥ 20 years of age
* Who give informed consent
* Confirmed diagnosis of RA (as defined by American College of Rheumatology revised 1987 criteria) and has ≥ 4 of the criteria listed below for ≥6 weeks before study enrollment
* Who self-pay or who are reimbursed by BNHI for abatacept treatment
* With latent TB or who are receiving anti-TB treatment (INH 300 mg, QD) 1 month prior to using abatacept and continuously up to a total of 9 months Willing to follow Taiwan Risk Management Plan guidelines as required by Taiwan health authorities
* Are being treated with abatacept or are abatacept treatment naïve and are initiating abatacept therapy

Exclusion Criteria:

* Pregnant or breast feeding
* With active TB
* HBsAg (+)and/or Anti-HCV(+) and/or HBV DNA(+)
* Have cancer (patients who were treated and have no sign of cancer for > 10 years can be included)
* Are allergic to abatacept
* Enrolled in other RA clinical studies

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital : Research based hospital centers, Teaching hospitals affiliated with medical schools, National/Regional medical centers and/or in which thought leaders are employed
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2014-08-06 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
The retention rate of abatacept therapy over 24 months in RA patients under real world clinical practice in Taiwan. | approximately 24 months
  Treatment retention rate is defined as the proportion of subjects who use abatacept for 24 months

SECONDARY OUTCOMES:
The retention rate (%) of abatacept therapy at 6, 9, 12, and 18 months in RA patients | at 6, 9, 12, 18, and 24months after study participation
The time to treatment discontinuation in RA patients treated with abatacept | at 6, 9, 12, 18, and 24months after study participation
  Treatment discontinuation is defined as patients who cease treatment for > 8 weeks
The proportion of patients achieving DAS28 ≤ 2.6, 2.6 < DAS28 ≤ 3.2, 3.2 < DAS28 ≤ 5.1, DAS> 5.1 at 6, 9, 12, 18, and 24months | at 6, 9, 12, 18, and 24months after study participation
The major reason for treatment discontinuation (eg, lack of efficacy, severe adverse drug reactions, switch from abatacept to another RA medication, financial issues, etc) at 6, 9, 12, 18, and 24 months | at 6, 9, 12, 18, and 24months after study participation
The demographic, clinical presentation, and disease management a composite measure of RA patients who are using abatacept (either formulation) or are abatacept naïve at Month 6, 9, 12, 18, and 24 | at 6, 9, 12, 18, and 24months after study participation

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Taipei, Taiwan

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm